CLINICAL TRIAL: NCT04124432
Title: Behavioral Pharmacology of Cannabis and Nicotine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB00220975; R21DA044377 (NIH)
Record Dates: First submitted 2019-10-10; First posted 2019-10-11 (Actual); Results first posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-03

CONDITIONS: Cannabis; Nicotine
MeSH Terms: conditions — Marijuana Abuse | interventions — nabiximols; Nicotine

STUDY DESIGN:
Intervention Model Description: All participants will complete all dose conditions (study arms) in a randomized order
Who Masked: Participant, Outcomes Assessor
Masking Description: placebo controlled, double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Active cannabis without nicotine (Experimental): Smoked cannabis containing 10mg THC + No nicotine/tobacco
  Interventions: Drug: Cannabis
- Active cannabis with own brand cigarettes (Experimental): Smoked cannabis containing 10mg THC + ad-libitum use of preferred brand cigarettes
  Interventions: Drug: Cannabis; Drug: Nicotine
- Active cannabis with low nicotine e-cigarette (Experimental): Smoked cannabis containing 10mg THC + ad-libitum use of low nicotine content E-Cig (3% nicotine JUUL)
  Interventions: Drug: Cannabis; Drug: Nicotine
- Active cannabis with high nicotine e-cigarette (Experimental): Smoked cannabis containing 10mg THC + ad-libitum use of high nicotine content E-Cig (5% nicotine JUUL)
  Interventions: Drug: Cannabis; Drug: Nicotine
- placebo cannabis with own brand cigarettes (Experimental): Smoked placebo cannabis + ad-libitum use of preferred brand cigarettes
  Interventions: Drug: Cannabis; Drug: Nicotine
- Placebo cannabis with low nicotine e-cigarette (Experimental): Smoked placebo cannabis + ad-libitum use of low nicotine content E-Cig (3% nicotine JUUL)
  Interventions: Drug: Cannabis; Drug: Nicotine
- Placebo cannabis with high nicotine e-cigarette (Experimental): Smoked placebo cannabis + ad-libitum use of high nicotine content E-Cig (5% nicotine JUUL)
  Interventions: Drug: Cannabis; Drug: Nicotine

INTERVENTIONS:
Drug: Cannabis — Cannabis will be smoked
Drug: Nicotine — Nicotine will be smoked or vaporized
  Arms: Active cannabis with high nicotine e-cigarette; Active cannabis with low nicotine e-cigarette; Active cannabis with own brand cigarettes; Placebo cannabis with high nicotine e-cigarette; Placebo cannabis with low nicotine e-cigarette; placebo cannabis with own brand cigarettes

SUMMARY:
This study will evaluate the individual and interactive pharmacokinetic and pharmacodynamic effects of smoked cannabis and nicotine.

DETAILED DESCRIPTION:
The proposed study will be conducted at the Johns Hopkins Behavioral Pharmacology Research Unit (BPRU). All participants will be healthy adult volunteers who are regular nicotine/tobacco users, and have prior experience with cannabis use. Participants will complete seven outpatient experimental test sessions (completed in a randomized order), under double-blind conditions in which participants will first self-administer smoked cannabis (either active or placebo), followed by nicotine (via a tobacco cigarette or an e-cigarette); there will also be one condition in which participants smoke active cannabis alone (without subsequent nicotine use). Nicotine self-administration will occur in an ad libitum fashion for 5 hours. Nicotine products will be the individual participant's preferred brand of cigarettes or the commercial pod-style e-cigarette the JUUL (pods will contain either 3% or 5% nicotine pods). Active cannabis will contain 10 mg tetrahydrocannabinol (THC) while placebo will contain 0 mg THC. During the ad libitum nicotine/tobacco-use period, various puffing behaviors (e.g., puff volume, puff duration, puff number, inter-puff-interval) will be measured using specialized equipment. Acute subjective effects of cannabis/nicotine, cannabis/nicotine withdrawal symptoms, craving, vital signs, and cognitive/psychomotor performance will also be assessed throughout the experimental sessions.

ELIGIBILITY:
Inclusion Criteria:

* Have provided written informed consent
* Be between the ages of 18 and 55
* Be in good general health based on a physical examination, medical history, vital signs, and screening urine and blood tests
* Test negative for drugs of abuse aside from cannabis (via urine sample) and alcohol (via breath sample) at the screening visit and upon arrival for each experimental session.
* Not be pregnant or nursing (if female). All females must have a negative serum pregnancy test at the screening visit and a negative urine pregnancy test at clinic admission.
* Have a body mass index (BMI) in the range of 18 to 36 kg/m2
* Blood pressure at screening visit does not exceed a systolic blood pressure (SBP) of 150 mmHg or a diastolic blood pressure (DBP) of 90 mmHg
* Have not donated blood in the prior 30 days.
* Report prior experience inhaling cannabis.
* Report using cannabis at least 5 times in the past year.
* Smoke ≥5 tobacco cigarettes per day on average in the past month.
* Use an e-cigarette at least 15 of the past 30 days.
* Have a breath carbon monoxide (CO) of >8ppm or urine cotinine >200ng/mL to confirm current nicotine use status.

Exclusion Criteria:

* Non-medical use of psychoactive drugs (aside from cannabis) other than, nicotine, alcohol, or caffeine in the month prior to the Screening Visit;
* History of or current evidence of significant medical or psychiatric illness which, in the opinion of the investigator or sponsor, will interfere with the study results or the safety of the subject.
* Use of an over-the-counter (OTC), systemic or topical drug(s), herbal supplement(s), or vitamin(s) within 14 days of experimental sessions; which, in the opinion of the investigator or sponsor, will interfere with the study results or the safety of the subject.
* Use of a prescription medication (with the exception of birth control prescriptions) within 14 days of experimental sessions; which, in the opinion of the investigator or sponsor, will interfere with the study results or the safety of the subject.
* History of clinically significant cardiac arrhythmias or vasospastic disease (e.g., Prinzmetal's angina).
* Enrolled in another clinical trial or have received any drug as part of a research study within 30 days prior to dosing.
* Epilepsy or a history of seizures.
* Individuals who have a recent history of traumatic brain injury diagnosed by CT/MRI and have current sequela from prior brain injury, as determined by the study physician
* Individuals with anemia.
* Prior history of allergic or serious adverse reaction to either cannabis or tobacco/nicotine.
* Average use of cannabis more than 2 times per week in the prior 3 months.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2023-07-24 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Vandrey, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cannabis With and Without Nicotine: This was a within-subjects, cross-over design in which all participants were exposed to all 7 conditions in a randomized order.
Period: Overall Study
Arm/Group | Cannabis With and Without Nicotine
Started | 26
THC + No Nicotine/Tobacco | 23
THC + Ad-libitum Use of Preferred Brand Cigarettes | 20
THC + Ad-libitum Use of Low Nicotine Content E-Cig (3% Nicotine JUUL) | 24
THC + Ad-libitum Use of High Nicotine Content E-Cig (5% Nicotine JUUL) | 22
Placebo Cannabis + Ad-libitum Use of Preferred Brand Cigarettes | 21
Placebo Cannabis + Ad-libitum Use of Low Nicotine Content E-Cig (3% Nicotine JUUL) | 22
Placebo Cannabis + Ad-libitum Use of High Nicotine Content E-Cig (5% Nicotine JUUL) | 21
Completed | 20
Not Completed | 6

BASELINE CHARACTERISTICS:
Population: We are reporting data for study completers. 20 participants completed the study.
Arm/Group | Cannabis With and Without Nicotine
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.47 (8.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Amount of Nicotine (mL of Smoke/Vapor) Inhaled
Description: Amount of nicotine used (determined by total volume (mL) of cigarette smoke or JUUL vapor inhaled) after cannabis exposure in each session.
Time Frame: 0-5 hours
Population: Represents study completers
Measure: Mean (Standard Deviation); unit: Volume in mL
Groups:
- Active Cannabis Without Nicotine: Smoked cannabis containing active THC + No nicotine/tobacco
  Cannabis: Cannabis will be smoked
- Active Cannabis With Own Brand Cigarettes: Smoked cannabis containing active THC + ad-libitum use of preferred brand cigarettes
  Cannabis: Cannabis will be smoked
  Nicotine: Nicotine will be smoked or vaporized
- Active Cannabis With Low Nicotine E-cigarette: Smoked cannabis containing active THC + ad-libitum use of low nicotine content E-Cig (3% nicotine JUUL)
  Cannabis: Cannabis will be smoked
  Nicotine: Nicotine will be smoked or vaporized
- Active Cannabis With High Nicotine E-cigarette: Smoked cannabis containing active THC + ad-libitum use of high nicotine content E-Cig (5% nicotine JUUL)
  Cannabis: Cannabis will be smoked
  Nicotine: Nicotine will be smoked or vaporized
Arm/Group | Active Cannabis Without Nicotine | Active Cannabis With Own Brand Cigarettes | Active Cannabis With Low Nicotine E-cigarette | Active Cannabis With High Nicotine E-cigarette | Placebo Cannabis With Own Brand Cigarettes | Placebo Cannabis With Low Nicotine E-cigarette | Placebo Cannabis With High Nicotine E-cigarette
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20 | 20
Volume in mL | 0 (0) | 489.0 (142.2) | 1814.0 (1064.0) | 1401.0 (1076.0) | 513.6 (247.2) | 1929.0 (2105.0) | 1390.0 (961.2)

2. Secondary Outcome: Mean Peak Change From Baseline Self-reported Drug Effect as Assessed by the Drug Effect Questionnaire (DEQ)
Description: Mean Peak Change From Baseline rating (0-100) of Drug Effect on the DEQ, with 0 being no effect and 100 being maximum effect.
Time Frame: 0-5 hours
Population: Represents study completers
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Cannabis Without Nicotine | Active Cannabis With Own Brand Cigarettes | Active Cannabis With Low Nicotine E-cigarette | Active Cannabis With High Nicotine E-cigarette | Placebo Cannabis With Own Brand Cigarettes | Placebo Cannabis With Low Nicotine E-cigarette | Placebo Cannabis With High Nicotine E-cigarette
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20 | 20
score on a scale | 46.9 (29.9) | 44.6 (30.1) | 47.5 (38.5) | 40.5 (36.5) | 21.4 (29.1) | 17.3 (26.1) | 9.4 (28.7)

3. Secondary Outcome: Mean Peak Change From Baseline Psychomotor Performance as Assessed by the Digit Symbol Substitution Task (DSST)
Description: Computerized version of Digit Symbol Substitution Task will be administered to assess psychomotor performance. Total correct trials in 90-seconds. Minimum score of 0 but no maximum score (higher scores indicate better performance).
Time Frame: 0-5 hours
Population: Represents study completers
Measure: Mean (Standard Deviation); unit: Total correct trials
Arm/Group | Active Cannabis Without Nicotine | Active Cannabis With Own Brand Cigarettes | Active Cannabis With Low Nicotine E-cigarette | Active Cannabis With High Nicotine E-cigarette | Placebo Cannabis With Own Brand Cigarettes | Placebo Cannabis With Low Nicotine E-cigarette | Placebo Cannabis With High Nicotine E-cigarette
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20 | 20
Total correct trials | -0.2 (7.0) | -0.5 (8.1) | -4.3 (6.9) | -3.3 (6.7) | 2.0 (5.9) | -3.6 (4.3) | -0.9 (8.1)

4. Secondary Outcome: Mean Peak Change From Baseline Working Memory Performance as Assessed by the Paced Auditory Serial Addition Task (PASAT)
Description: Computerized version of Paced Auditory Serial Addition Task will be administered to assess working memory performance. Total correct trials out of 90 recorded is primary outcome (higher scores indicate better performance).
Time Frame: 0-5 hours
Population: Represents study completers
Measure: Mean (Standard Deviation); unit: Total correct trials
Arm/Group | Active Cannabis Without Nicotine | Active Cannabis With Own Brand Cigarettes | Active Cannabis With Low Nicotine E-cigarette | Active Cannabis With High Nicotine E-cigarette | Placebo Cannabis With Own Brand Cigarettes | Placebo Cannabis With Low Nicotine E-cigarette | Placebo Cannabis With High Nicotine E-cigarette
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20 | 20
Total correct trials | -3.8 (9.1) | 0.9 (15.4) | -9.8 (12.0) | -1.2 (11.1) | 5.3 (21.6) | -5.7 (9.6) | -6.9 (9.2)

5. Secondary Outcome: Mean Peak Change From Baseline Behavioral Task Performance as Assessed by the DRUID App
Description: Behavioral task performance will be assessed with the DRUID app's Global impairment score (range 0-100), where lower scores indicate better performance.
Time Frame: 0-5 hours
Population: Represents study completers
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Cannabis Without Nicotine | Active Cannabis With Own Brand Cigarettes | Active Cannabis With Low Nicotine E-cigarette | Active Cannabis With High Nicotine E-cigarette | Placebo Cannabis With Own Brand Cigarettes | Placebo Cannabis With Low Nicotine E-cigarette | Placebo Cannabis With High Nicotine E-cigarette
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20 | 20
score on a scale | 4.3 (12.0) | -0.3 (7.4) | 3.0 (7.4) | 2.1 (6.4) | -1.3 (10.3) | -4.8 (13.6) | 0.3 (6.7)

6. Secondary Outcome: Mean Peak Change From Baseline Tobacco Craving as Assessed by the Tobacco Craving Questionnaire
Description: Mean peak change from baseline rating (0-100) of "Craving" with 0 being no craving and 100 being maximum craving.
Time Frame: 0-5 hours
Population: Represents study completers
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Cannabis Without Nicotine | Active Cannabis With Own Brand Cigarettes | Active Cannabis With Low Nicotine E-cigarette | Active Cannabis With High Nicotine E-cigarette | Placebo Cannabis With Own Brand Cigarettes | Placebo Cannabis With Low Nicotine E-cigarette | Placebo Cannabis With High Nicotine E-cigarette
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20 | 20
score on a scale | 0.6 (2.6) | -0.8 (2.4) | 0.0 (2.7) | -0.2 (3.0) | -0.2 (2.3) | 0.6 (1.8) | 0.8 (3.2)

7. Secondary Outcome: Mean Peak Change From Baseline Cannabis Craving as Assessed by the Cannabis Craving Questionnaire
Description: Mean peak change from baseline rating (0-100) of "Craving" with 0 being no craving and 100 being maximum craving
Time Frame: 0-5 hours
Population: Represents study completers
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Cannabis Without Nicotine | Active Cannabis With Own Brand Cigarettes | Active Cannabis With Low Nicotine E-cigarette | Active Cannabis With High Nicotine E-cigarette | Placebo Cannabis With Own Brand Cigarettes | Placebo Cannabis With Low Nicotine E-cigarette | Placebo Cannabis With High Nicotine E-cigarette
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20 | 20
score on a scale | -1.9 (2.5) | -1.6 (2.2) | -1.7 (2.6) | -2.6 (1.7) | -1.0 (2.1) | -0.9 (1.5) | -0.9 (2.4)

ADVERSE EVENTS:
Time Frame: 0-5 hours
Description: International Council for Harmonization (ICH) guidelines are followed for Adverse Event (AE) reporting, as AEs occur they are documented.
Arm/Group | Active Cannabis Without Nicotine | Active Cannabis With Own Brand Cigarettes | Active Cannabis With Low Nicotine E-cigarette | Active Cannabis With High Nicotine E-cigarette | Placebo Cannabis With Own Brand Cigarettes | Placebo Cannabis With Low Nicotine E-cigarette | Placebo Cannabis With High Nicotine E-cigarette
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/20 | 0/24 | 0/22 | 0/21 | 0/22 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/20 | 0/24 | 0/22 | 0/21 | 0/22 | 0/21
Other Adverse Events (participants affected / at risk) | 0/23 | 0/20 | 1/24 | 0/22 | 1/21 | 0/22 | 0/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Cannabis Without Nicotine (N=23) | Active Cannabis With Own Brand Cigarettes (N=20) | Active Cannabis With Low Nicotine E-cigarette (N=24) | Active Cannabis With High Nicotine E-cigarette (N=22) | Placebo Cannabis With Own Brand Cigarettes (N=21) | Placebo Cannabis With Low Nicotine E-cigarette (N=22) | Placebo Cannabis With High Nicotine E-cigarette (N=21)
Vomitting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-15): https://cdn.clinicaltrials.gov/large-docs/32/NCT04124432/Prot_SAP_000.pdf